CLINICAL TRIAL: NCT06794112
Title: Optimal Bowel Preparation in Geriatric Patients With a Instructional Animation Video Before Colonoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Hilmi Bozkurt, Associate Professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2024/1269
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Bowel Preparation Before Colonoscopy; Geriatric Patient; Instructional Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animation video group (Experimental): Patients will receive standard written instructions and will additionally watch an animated training video
  Interventions: Other: Animated Educational Video; Other: Written Instructions
- Written instructions only (Standard care) group (Active Comparator): Patients will only receive standardised written instructions
  Interventions: Other: Written Instructions

INTERVENTIONS:
Other: Animated Educational Video — Both arms will receive standard care (written instructions), with the experimental arm receiving an additional animated video intervention.
  Arms: Animation video group
Other: Written Instructions — Standard written instructions for bowel preparation before colonoscopy

SUMMARY:
Our study presents an innovative educational approach combining visual and auditory elements, targeting the specific needs of the geriatric population. Generally, before colonoscopy, participants are given a written instruction describing the standard bowel preparation with the use of laxatives and enemas. In our study, in addition to this written instruction, the investigators aimed to support the bowel preparation procedure with visual training by using an animated video. The use of animated video has the potential to present complex medical instructions in a simple and understandable format. This approach is especially designed for elderly participants who have limited literacy skills or have difficulty in following written instructions. In addition, it was aimed to reduce the anxiety of the participants before the colonoscopy procedure and to increase patient compliance.

DETAILED DESCRIPTION:
Colonoscopy is a critical screening method for early detection and prevention of colorectal cancer. However, the success of the procedure largely depends on the quality of bowel preparation. Inadequate bowel preparation may lead to repeated procedures, increased costs, potentially delayed diagnoses and associated poor prognosis. This problem is more prominent especially in the geriatric population over 60 years of age. With the animated video, the investigators aim to improve bowel cleansing before colonoscopy by providing visual and auditory training to participants and/or their carers. This project will both contribute to the improvement of colonoscopy preparation protocols for the geriatric population and potentially provide a model that can be adapted to other age groups.

Animation training video was created collaboratively by Mersin University Faculty of Medicine Department of General Surgery and Mersin University Graphic Arts Department.

The Boston Bowel Preparation Scale (BBPS) is a scoring system designed to assess bowel cleansing during colonoscopy. It provides a standardised, reliable measure to improve the quality and outcomes of colonoscopy procedures. While there are many different scales to measure bowel preparation, the BBPS was selected for use in the study as it is considered to be the most comprehensively validated bowel preparation scale. The BBPS is a 10-point scale that assesses bowel readiness. It assesses three segments of the colon (right, transverse and left) with scores ranging from 0 to 3 for each segment, leading to a total score of 0 to 9.

Using this scale, the investigators tried to determine whether there would be a difference in terms of bowel preparation between participants who watched an animated video and participants who were given standard instructions.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Indication for colonoscopy
* Volunteering to participate in the study
* Preparing for colonoscopy for the first time
* No history of previous operations on the small intestine and colon
* No diagnosed bowel disease
* Language proficiency to watch the animation
* Full understanding of visual and auditory messages

Exclusion Criteria:

* Previous colonoscopy experience
* History of previous small bowel and colon surgery
* Diagnosis of inflammatory bowel disease
* Presence of toxic colon and/or megacolon
* The presence of a mass in the intestine that does not allow colonoscopy to pass
* Unwillingness to participate in the study
* Lack of language proficiency
* Lack of ability to understand visual and auditory messages

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Bowel Preparation | During colonoscopy procedure
  The primary outcome measure of this study is the quality of bowel preparation, which will be assessed using the Boston Bowel Preparation Scale (BBPS). This validated scale will be used to evaluate the cleanliness of each colonic segment during colonoscopy. The BBPS assigns a score of 0 to 3 for each of the three segments of the colon (right colon, transverse colon, and left colon), resulting in a total score ranging from 0 to 9. Adequate bowel preparation will be defined as a total BBPS score ≥ 6 with all segment scores ≥ 2. The assessment will be performed by endoscopists who are blinded to the patient's group allocation to minimize bias. This standardized evaluation will provide an objective measure of the effectiveness of our video-based educational intervention compared to standard written instructions in achieving optimal bowel preparation in the geriatric population.

SECONDARY OUTCOMES:
colonoscopy completion rate | During colonoscopy procedure
  This will be documented by the endoscopist during the procedure and recorded as a binary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Simge Tuna, Study Chair — Mersin University
Locations (1):
- Mersin University Faculty of Medicine, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ye Z, Chen J, Xuan Z, Gao M, Yang H. Educational video improves bowel preparation in patients undergoing colonoscopy: a systematic review and meta-analysis. Ann Palliat Med. 2020 May;9(3):671-680. doi: 10.21037/apm.2020.03.33. Epub 2020 Apr 13. PMID 32312062
- [Background] Ho LH, Montealegre JR, Al-Arabi S, Jibaja-Weiss ML, Suarez MG. Impact of Colonoscopy Preparation Video on Boston Bowel Preparation Scale Score. Gastroenterol Nurs. 2019 May/Jun;42(3):251-258. doi: 10.1097/SGA.0000000000000391. PMID 31145249
- [Background] Hayat U, Lee PJ, Lopez R, Vargo JJ, Rizk MK. Online Educational Video Improves Bowel Preparation and Reduces the Need for Repeat Colonoscopy Within Three Years. Am J Med. 2016 Nov;129(11):1219.e1-1219.e9. doi: 10.1016/j.amjmed.2016.06.011. Epub 2016 Jul 6. PMID 27393880